CLINICAL TRIAL: NCT04536766
Title: Impact of Bed Provision and Enhanced Sleep Health Education on Sleep in Socio-economically Disadvantaged Children
Brief Title: Impact of Bed Provision and Sleep Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Joseph's University, Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01
Record Dates: First submitted 2020-08-16; First posted 2020-09-03 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-04

CONDITIONS: Sleep Disturbance; Sleep Deprivation; Sleep; Insomnia
MeSH Terms: conditions — Parasomnias; Sleep Deprivation; Sleep Initiation and Maintenance Disorders | interventions — Beds

STUDY DESIGN:
Intervention Model Description: 100 Caregiver-child dyads (children ages 8-12 years) will be recruited from the Beds for Kids program.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Sleep Health Education (Experimental): 50 families will be randomly assigned to receive sleep health education delivered in two telephone sessions by Beds for Kids staff members, in addition to receiving the standard Beds for Kids program (bed, bedding, written sleep education materials). The first session will occur approximately 2-3 days before bed delivery. The second 15-20-minute session will occur approximately one week following bed delivery. Sleep health education training and supervision of Beds for Kids staff members will be provided by board-certified Behavioral Sleep Medicine providers. Sleep health information will be manualized and will consist of evidence-based pediatric sleep health behaviors: ensuring adequate sleep duration, developing a bedtime routine, keeping a regular sleep schedule, avoiding caffeine, and eliminating electronics in the bedroom and at bedtime. The enhanced sleep health intervention sessions will also include individualized problem-solving and tailoring to meet the family's needs.
  Interventions: Behavioral: Enhanced Sleep Health Education
- Beds for Kids Standard Program (Active Comparator): 50 families will be randomly assigned to the standard Beds for Kids program, which includes a bed, bedding, and written sleep education materials.
  Interventions: Behavioral: Beds for Kids Standard Program

INTERVENTIONS:
Behavioral: Enhanced Sleep Health Education — The intervention comprehensively addresses poor sleep health behaviors. Personalized sleep health education will be delivered in two telephone sessions by Beds for Kids staff members. Sleep health information will consist of the following evidence-based pediatric sleep health behaviors: ensuring adequate sleep duration, developing a family bedtime routine, keeping a regular sleep schedule, avoiding caffeine, and eliminating electronics in the bedroom and at bedtime. The enhanced sleep health intervention sessions will also include individualized problem-solving and tailoring to meet the family's needs. Personalization will be accomplished via direct questions to families during the education phone call related to their own barriers to achieving healthy sleep habits and goals for optimal sleep.
  Arms: Enhanced Sleep Health Education
Behavioral: Beds for Kids Standard Program — The Beds for Kids program provides beds, bedding, and written healthy sleep education to families living at or below 100% of the federal poverty line and without an individual child bed to sleep in.
  Arms: Beds for Kids Standard Program

SUMMARY:
Investigators will recruit up to 100 families (children aged 8-12 years and their primary caregivers) from the Philadelphia-area Beds for Kids charity program, which provides beds, bedding, and sleep education to lower-socioeconomic status (SES) children. The primary objective of this randomized controlled trial is to determine whether bed provision combined with provider-delivered sleep health education can improve sleep in children participating in the Beds for Kids program.

DETAILED DESCRIPTION:
Insufficient and poor-quality sleep impacts more than half of school-aged children, and is associated with significant impairments in child neurocognitive, academic, behavioral, and physical health functioning. Lower socioeconomic status (SES) children are at increased risk for poor sleep. Compared to their higher-SES peers, lower-SES youth tend to obtain less sleep overall and experience worse sleep quality. Many children of lower-SES also may live in noisy or high-violence neighborhoods and in overcrowded homes that lack a child bed or other designated child sleep space. These environmental factors may perpetuate SES-related health disparities in child sleep duration, quality, and poor sleep health behaviors (i.e., bedroom electronics). Although there is a robust evidence-base for treating childhood sleep problems, there is a paucity of sleep intervention research focused on lower-SES children.

Beds for Kids is a Philadelphia-area program that is part of the larger volunteer organization, One House at a Time, that provides lower-SES children with beds, bedding, and a sleep education brochure. To qualify for program participation, youth must be: (1) between the ages of 2 and 20 years, (2) living without an individual bed (e.g., sleeping on the floor, on a sofa, or crowded into one bed with family members), and (3) living in a household whose income is at or below 100 percent of the United States poverty threshold. The program accepts referrals from area social service agencies in the greater Philadelphia area.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver participant is the parent or legal guardian of the child participant.
* Caregiver/legal guardian is 18 years of age.
* Child between 8 and 12 years of age.
* English-speaking

Exclusion Criteria:

* Caregiver is not parent or legal guardian of child participant.
* Presence of a diagnosed child neurodevelopmental (e.g., autism spectrum disorder, Trisomy 21) or chronic medical condition (e.g., sickle cell disease, cancer) in which the disorder or treatment of the disorder impact sleep.
* Caregivers/guardians or subjects who, in the opinion of the Investigator, may be non- compliant with study schedules or procedures.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2020-10-24 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Treatment acceptability: Treatment Evaluation Inventory-Short Form | 2 months
  Caregivers randomized to the enhanced sleep health education arm will complete the Treatment Evaluation Inventory-Short Form, a widely used measure of treatment acceptability that has been adapted for the purposes of the Beds for Kids intervention. Caregivers will complete an electronic survey with questions related to aspects of the intervention including perceived efficacy/helpfulness and acceptability of the intervention. Seven items will be rated on a 5-point Likert scale from 1 'strongly disagree' and to 5 'strongly agree' with total scores ranging from 1 to 35 (higher scores denoting higher acceptability). In addition, the percent of participants who indicate they "agree" or "strongly agree" for each of the 4 items (acceptability of measures) and 3 items (helpfulness) will be reported.
Sleep health-related behaviors | 2 months
  The Pediatric Sleep Practices Questionnaire is a 7 item measure related to sleep health-related practices, including bedtime routine consistency, the use of electronics prior to bedtime, sleep schedule regularity, and parental presence at bedtime, resulting in three subscales: total sleep timing (range 0-4), total routines/consistency (range 0-6), and total sleep environment (range 0-6). Two additional subscales include technology usage before bed (range 0-4) and the child's need for someone to fall asleep with them (range 0-2). Total scores range from 0 to 22. Higher scores denote poorer sleep practices.
Sleep outcomes | 2 months
  Children and their caregivers will report on child sleep disturbance and sleep-related impairments, using the reliable and valid Patient-Reported Outcomes Measurement Information System (PROMIS) self-and caregiver-proxy-report scales for pediatric sleep. To measure sleep disturbance, the PROMIS Parent Proxy Sleep Disturbance - Short Form 8a and the PROMIS Pediatric Sleep Disturbance - Short Form 8a will be completed. For the measurement of impairments of daily function related to lack of sleep, the PROMIS Parent Proxy Sleep-Related Impairment - Short Form 8a and the PROMIS Pediatric Sleep-Related Impairment - Short Form 8a will be completed.
  Items on all four assessments are rated on a 5-point Likert scale from 1 'never' to 5 'always,' with total sum scores for each measure ranging from 1 to 40 (higher scores denoting greater sleep disturbance or impairment). Scores will be converted into normative-based T-scores.

SECONDARY OUTCOMES:
Family engagement | 12 months
  Family engagement will be based on percent completion of sleep education phone calls (possible range = 0-100%) for the intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph's University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Allen SL, Howlett MD, Coulombe JA, Corkum PV. ABCs of SLEEPING: A review of the evidence behind pediatric sleep practice recommendations. Sleep Med Rev. 2016 Oct;29:1-14. doi: 10.1016/j.smrv.2015.08.006. Epub 2015 Sep 1. PMID 26551999
- [Background] Astill RG, Van der Heijden KB, Van Ijzendoorn MH, Van Someren EJ. Sleep, cognition, and behavioral problems in school-age children: a century of research meta-analyzed. Psychol Bull. 2012 Nov;138(6):1109-38. doi: 10.1037/a0028204. Epub 2012 Apr 30. PMID 22545685
- [Background] Buxton OM, Chang AM, Spilsbury JC, Bos T, Emsellem H, Knutson KL. Sleep in the modern family: protective family routines for child and adolescent sleep. Sleep Health. 2015 May 1;1(1):15-27. doi: 10.1016/j.sleh.2014.12.002. PMID 26779564
- [Background] Bagley EJ, Kelly RJ, Buckhalt JA, El-Sheikh M. What keeps low-SES children from sleeping well: the role of presleep worries and sleep environment. Sleep Med. 2015 Apr;16(4):496-502. doi: 10.1016/j.sleep.2014.10.008. Epub 2014 Dec 16. PMID 25701537
- [Background] Dewald JF, Meijer AM, Oort FJ, Kerkhof GA, Bogels SM. The influence of sleep quality, sleep duration and sleepiness on school performance in children and adolescents: A meta-analytic review. Sleep Med Rev. 2010 Jun;14(3):179-89. doi: 10.1016/j.smrv.2009.10.004. Epub 2010 Jan 21. PMID 20093054
- [Background] El-Sheikh M, Bagley EJ, Keiley M, Elmore-Staton L, Chen E, Buckhalt JA. Economic adversity and children's sleep problems: multiple indicators and moderation of effects. Health Psychol. 2013 Aug;32(8):849-59. doi: 10.1037/a0030413. Epub 2012 Nov 12. PMID 23148451
- [Background] Forrest CB, Meltzer LJ, Marcus CL, de la Motte A, Kratchman A, Buysse DJ, Pilkonis PA, Becker BD, Bevans KB. Development and validation of the PROMIS Pediatric Sleep Disturbance and Sleep-Related Impairment item banks. Sleep. 2018 Jun 1;41(6). doi: 10.1093/sleep/zsy054. PMID 29546286
- [Background] Jarrin DC, McGrath JJ, Quon EC. Objective and subjective socioeconomic gradients exist for sleep in children and adolescents. Health Psychol. 2014 Mar;33(3):301-5. doi: 10.1037/a0032924. Epub 2013 Jun 3. PMID 23730721
- [Background] Kelley ML, Heffer RW, Gresham FM, Elliott SN. Development of a modified treatment evaluation inventory. Journal of Psychopathology and Behavioral Assessment. 1989;11(3):235-247.
- [Background] Miller MA, Kruisbrink M, Wallace J, Ji C, Cappuccio FP. Sleep duration and incidence of obesity in infants, children, and adolescents: a systematic review and meta-analysis of prospective studies. Sleep. 2018 Apr 1;41(4). doi: 10.1093/sleep/zsy018. PMID 29401314
- [Background] Mindell JA, Sedmak R, Boyle JT, Butler R, Williamson AA. Sleep Well!: A Pilot Study of an Education Campaign to Improve Sleep of Socioeconomically Disadvantaged Children. J Clin Sleep Med. 2016 Dec 15;12(12):1593-1599. doi: 10.5664/jcsm.6338. PMID 27655459